CLINICAL TRIAL: NCT06182605
Title: Multifunctional Cataract Surgery Assistive Instruments Used in Cataract Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0370
Record Dates: First submitted 2023-12-07; First posted 2023-12-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-functional instruments (Experimental): Patients undergoing cataract with lens subluxation surgery with Multifunctional cataract-assisted retractor
  Interventions: Device: multifunctional instruments
- Traditional instruments (Active Comparator): Patients undergoing cataract with lens subluxation surgery with traditional capsule retractor
  Interventions: Device: traditional instruments

INTERVENTIONS:
Device: multifunctional instruments — Ophthalmic retractors can be used to lift the lens during surgery to assist in lens sucking or resection; Intraoperative injection of reagent, which has the advantage of retractable, micro-incision. Ophthalmic hooks can be used to secure support capsular bags; auxiliary cleavage; polishing capsule; Viscoelastic agent is injected as needed. The front end of the membranous cataract scissor is a capsular tearing forceps, and the capsule tearing and capsule scissors can be flexibly switched. All three instruments have the functions of two or three traditional instruments, which can be designed to reduce the number of times the instruments enter and exit the incision during surgery, improve surgical efficiency,
  Other Names: A set of available instruments including ophthalmic retractor, ophthalmic hook and membranous cataract scissors,
  Arms: Multi-functional instruments
Device: traditional instruments — traditional Cataract-assisted instruments for cataract operation.Puncture knives, microscissors, microscopic forceps, nucleus hooks, lens graft forceps, are used to cut the cornea, assist in removing the cloudy lens, suturing wounds.
  Other Names: commonly used instruments for cataract surgery
  Arms: Traditional instruments

SUMMARY:
In order to better cope with complex situations of cataract surgery, we designed and improved a new set of multi-functional cataract surgery auxiliary devices, including ophthalmic surgery auxiliary hooks, eye retractor hooks and membranous cataract scissors. Their common feature is that they have the function of 2-3 traditional surgical instruments, which can be switched in operations, reducing the replacement of different surgical instruments, lowing the number of surgical instruments in and out of the incision, reducing trauma and improving surgical efficiency. The purpose of this multi-center prospective clinical study is to verify the advantages of this new group of multifunctional devices and further summarize the experience and improvement by comparing the safety and effectiveness of traditional cataract surgical instruments combined with new multifunctional cataract assisted surgical instruments and traditional cataract surgical instruments alone.

DETAILED DESCRIPTION:
Cataract is the number one cause of blindness, and the main treatment method is surgery to remove the cloudy lens and install an intraocular lens. The operation relies on ophthalmic micromanipulative instruments, but in complex cases such as abnormal lens capsule, ocular trauma, etc., the difficulty of surgery increases, so that conventional instruments are often unable to complete the operation well. In order to better cope with these complex situations, we designed and improved a new set of multi-functional cataract surgery auxiliary devices, including ophthalmic surgery auxiliary hooks, eye retractor hooks and membranous cataract scissors, which have obtained utility model patents and first-class medical device filings. Their common feature is that they have the function of 2-3 traditional surgical instruments, which can be switched intraoperatively, reduce the replacement of different surgical instruments, reduce the number of surgical instruments in and out of the incision, reduce trauma and improve surgical efficiency. The purpose of this multi-center prospective clinical study is to verify the advantages of this new group of multifunctional devices and further summarize the experience and improvement by comparing the safety and effectiveness of traditional cataract surgical instruments combined with new multifunctional cataract assisted surgical instruments and traditional cataract surgical instruments alone.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of cataract Patients need to undergo cataract surgery

Exclusion Criteria:

- Active intraocular inflammation The intraocular pressure (IOP) was higher than 25 mmHg The endothelial cell count (ECC) was less than 1,200 cells/mm2 Combined with other eye diseases Combined with other serious systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Successful implantation rate of intraocular lens | through study completion, an average of 1 year
  implantation rate of intraocular lens with different instrument

SECONDARY OUTCOMES:
Visual function | 1day postoperation，1 week，1 month， 3month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart Best corrected visual acuity (BCVA) measured using a decimal chart
intraocular pressure | 1 day, 1 week, 1 month, and 3 month postoperation
  intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No